CLINICAL TRIAL: NCT01439165
Title: Safety and Immunogenicity in Adults of Revaccination With Adacel® Vaccine 10 Years After a Previous Dose
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Td537; U1111-1117-7012 (Other: WHO)
Record Dates: First submitted 2011-09-20; First posted 2011-09-23 (Estimated); Results first posted 2017-10-09 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-03

CONDITIONS: Tetanus; Diphtheria; Pertussis; Whooping Cough
Keywords: Adacel vaccine; Tetanus; Diphtheria; whooping cough
MeSH Terms: conditions — Tetanus; Diphtheria; Whooping Cough | interventions — Tetanus Toxoid; Diphtheria Toxoid; Pertussis Vaccine; adacel; Diphtheria-Tetanus Vaccine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adacel® Vaccine Group (Experimental): Participants randomized to receive a repeat dose of Tetanus Toxoid, Diphtheria Toxoid and Pertussis Vaccine (Adacel®)
  Interventions: Biological: Tetanus Toxoid, Diphtheria Toxoid and Pertussis Vaccine
- Td Adsorbed Vaccine Group (Active Comparator): Participants randomized to receive Subjects randomized to receive a Tetanus and Diphtheria Toxoids Adsorbed For Adult Use (TENIVAC) vaccine.
  Interventions: Biological: Tetanus and Diphtheria Toxoids Adsorbed For Adult Use

INTERVENTIONS:
Biological: Tetanus Toxoid, Diphtheria Toxoid and Pertussis Vaccine — 0.5 mL, Intramuscular
  Other Names: Adacel®
  Arms: Adacel® Vaccine Group
Biological: Tetanus and Diphtheria Toxoids Adsorbed For Adult Use — 0.5 mL, Intramuscular
  Other Names: TENIVAC
  Arms: Td Adsorbed Vaccine Group

SUMMARY:
The purpose of this study is to describe the safety and immunogenicity of repeat administration of Adacel vaccine approximately 10 years following initial administration of the vaccine. Antibody levels prior to revaccination will also be used to characterize antibody persistence following initial vaccination 10 years earlier.

Primary Objectives:

* To compare seroprotection rates against tetanus and diphtheria induced by Adacel vaccine to those induced by Td Adsorbed vaccine.
* To compare booster response rates against tetanus and diphtheria induced by Adacel vaccine to those induced by Td Adsorbed vaccine.
* To compare anti-pertussis geometric mean antibody concentrations (GMCs) induced by Adacel vaccine to the GMCs induced by Daptacel® vaccine given to infants.

Secondary Objectives:

* To describe the rates of immediate reactions, solicited reactions, unsolicited adverse events (AEs), and serious adverse events (SAEs) following vaccination with Adacel or Td Adsorbed vaccine.
* To describe booster response rates for pertussis antigens following revaccination with Adacel vaccine.

DETAILED DESCRIPTION:
Healthy adults < 65 years of age who received Adacel vaccine 10 years previously will be randomized to receive either Adacel or TENIVAC (Td Adsorbed) vaccine. They will be assessed for immunogenicity at baseline and post-vaccination. Safety data will be collected for 6 months following vaccination.

ELIGIBILITY:
Inclusion criteria:

* Subject is ≥ 18 to < 65 years of age at the time of vaccination.
* Received Adacel vaccine no less than 9 and no more than 11 years previously.
* Informed consent form has been signed and dated.
* Subject is able to attend all scheduled visits and to comply with all trial procedures.

Exclusion criteria:

* Subject is pregnant, or lactating, or of child bearing potential without using an effective method of contraception or not practicing abstinence for at least 4 weeks prior to vaccination and until at least 4 weeks after vaccination. Females who are pre-menarche or post-menopausal for at least one year, or surgically sterile will not be excluded.
* Any condition that, in the opinion of the Investigator, would pose a health risk to the participant or interfere with the evaluation of the vaccine.
* Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with trial conduct or completion.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* Known or suspected receipt of tetanus toxoid (T), tetanus and diphtheria toxoids (Td), or tetanus and diphtheria toxoids and acellular pertussis (Tdap) vaccine since receipt of the qualifying dose of Adacel vaccine described in Inclusion Criterion #2.
* A personal history of physician-diagnosed or laboratory-confirmed pertussis disease within the last 10 years.
* A previous severe reaction to pertussis, diphtheria or tetanus vaccine including immediate anaphylaxis, encephalopathy within 7 days or seizure within 3 days of receiving the vaccine.
* Receipt of immune globulins, blood or blood-derived products in the past 3 months.
* Suspected or known hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine used in the trial or to a vaccine containing any of the same substances.
* Receipt of any vaccine within 30 days before receiving study vaccine, or plans to receive another vaccine before the 2nd visit; except that influenza vaccine may have been received between 30 and 15 days (but no less than 15 days) before receiving study vaccine.
* Participation in another interventional clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 30 days preceding the first study vaccination or during the course of the study, at the discretion of the Sponsor.
* Seropositivity for Human Immunodeficiency Virus (HIV), Hepatitis B, or Hepatitis C, as reported by the subject.
* Laboratory-confirmed thrombocytopenia, which may be a contraindication for IM vaccination, at the discretion of the Investigator.
* Bleeding disorder or receipt of anticoagulants in the 3 weeks preceding inclusion, which may be a contraindication for intramuscular (IM) vaccination, at the discretion of the Investigator.
* Personal history of Guillain-Barré syndrome.
* Moderate or severe acute illness/infection (according to Investigator judgment) or febrile illness (temperature ≥ 38.0°C [≥ 100.4°F]) on the day of vaccination. A prospective subject should not be enrolled in the study until the condition has resolved or the febrile event has subsided.
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study.
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
* Current alcohol or drug use that, in the opinion of the Investigator, might interfere with the ability to comply with trial procedures.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1330 (Actual)
Dates: Start 2011-11; Primary Completion 2015-12 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (33):
- United States (31):
  - Huntsville, Alabama
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - San Diego, California
  - Boulder, Colorado
  - Marietta, Georgia
  - Woodstock, Georgia
  - Peoria, Illinois
  - Mishawaka, Indiana
  - Louisville, Kentucky
  - Rockville, Maryland
  - Woburn, Massachusetts
  - Columbia, Missouri
  - St Louis, Missouri
  - Albuquerque, New Mexico
  - Brooklyn, New York
  - Ithaca, New York
  - Rochester, New York
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Clairton, Pennsylvania
  - Hershey, Pennsylvania
  - Latrobe, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Syracuse, Utah
  - Virginia Beach, Virginia
  - Vancouver, Washington
  - Chippewa Falls, Wisconsin
  - Marshfield, Wisconsin
- Canada (2):
  - Harbour Grace, Newfoundland and Labrador
  - St. John's, Newfoundland and Labrador

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Result] Halperin SA, Donovan C, Marshall GS, Pool V, Decker MD, Johnson DR, Greenberg DP; Tdap Booster Investigators. Randomized Controlled Trial of the Safety and Immunogenicity of Revaccination With Tetanus-Diphtheria-Acellular Pertussis Vaccine (Tdap) in Adults 10 Years After a Previous Dose. J Pediatric Infect Dis Soc. 2019 May 11;8(2):105-114. doi: 10.1093/jpids/pix113. PMID 29438562
- [Derived] Pool V, Tomovici A, Johnson DR, Greenberg DP, Decker MD. Humoral immunity 10 years after booster immunization with an adolescent and adult formulation combined tetanus, diphtheria, and 5-component acellular pertussis vaccine in the USA. Vaccine. 2018 Apr 19;36(17):2282-2287. doi: 10.1016/j.vaccine.2018.03.029. Epub 2018 Mar 21. PMID 29573876

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 30 November 2011 to 13 August 2015 at 31 clinic sites in the United States and 2 clinic sites in Canada.
Pre-assignment Details: A total of 1330 participants who met all inclusion criteria and no exclusion criteria were randomized; 1327 participants were vaccinated.
Groups:
- Adacel Vaccine: Healthy adults <65 years of age who received Adacel 10 years ago received a repeat dose of Adacel vaccine.
- Td Adsorbed Vaccine: Healthy adults <65 years of age who received Adacel 10 years ago received TENIVAC® (Td Adsorbed vaccine).
Period: Overall Study
Arm/Group | Adacel Vaccine | Td Adsorbed Vaccine
Started | 1002 | 328
Completed | 981 | 326
Not Completed | 21 | 2
Not completed — Protocol Violation | 3 | 0
Not completed — Lost to Follow-up | 11 | 1
Not completed — Withdrawal by Subject | 7 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adacel Vaccine | Td Adsorbed Vaccine | Total
Number analyzed (Participants) | 1002 | 328 | 1330
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1002 | 328 | 1330
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Age Continuous | 28.9 (10.0) | 29.2 (10.6) | 29 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 646 | 212 | 858
  Male | 356 | 116 | 472
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 270 | 84 | 354
  Canada | 732 | 244 | 976

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Diphtheria and Tetanus Seroprotection
Description: Anti-Diphtheria antibodies were assessed by a toxin neutralization test. Anti-Tetanus antibodies were assessed using an enzyme-linked immunosorbent assay. Seroprotection was defined as the following: Anti-Diphtheria and Anti-Tetanus ≥ 0.1 IU/mL.
Time Frame: 1 month post-booster vaccination
Population: Seroprotection was assessed in the Per Protocol Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | Adacel Vaccine | Td Adsorbed Vaccine
Number analyzed (Participants) | 948 | 317
Percentage of participants
  Tetanus | 100.0 | 100.0
  Diphtheria | 99.8 | 99.4
Statistical Analysis 1: Comparison: Adacel Vaccine vs Td Adsorbed Vaccine; Comparison of anti-tetanus seroprotection rate between the two groups; Test type: Non-Inferiority — Non-inferiority concluded if the lower limit of the 2-sided 95% Confidence Interval (CI) of the difference of seroprotection rates between groups is > -10%; Difference (%) in Adacel-Td Adsorbed = 0.0, 95% CI 2-sided [-0.4 to 1.2]
Statistical Analysis 2: Comparison: Adacel Vaccine vs Td Adsorbed Vaccine; Comparison of anti-diphtheria seroprotection rates between the two groups; Test type: Non-Inferiority — Non-inferiority concluded if the lower limit of the 2-sided 95% CI of the difference of seroprotection rates between groups is > -10%; Difference (%) in Adacel-Td Adsorbed = 0.42, 95% CI 2-sided [-0.3 to 2.1]

2. Primary Outcome: Percentage of Participants With Diphtheria and Tetanus Booster Response
Description: Anti-Diphtheria antibodies were assessed by a toxin neutralization test. Anti-Tetanus antibodies were assessed using an enzyme-linked immunosorbent assay. A booster response was defined as a 4-fold increase in pre- to post-vaccination antibody concentrations for subjects with pre-vaccination antibody concentrations ≤2.56 IU/mL for diphtheria and ≤ 2.7 IU/mL for tetanus. If the pre vaccination antibody concentrations were > 2.56 IU/mL for diphtheria and > 2.7 IU/mL for tetanus, then a 2-fold increase in response rate was defined as a booster response.
Time Frame: 1 month post-booster vaccination
Population: Booster response rates were assessed in the Per Protocol Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | Adacel Vaccine | Td Adsorbed Vaccine
Number analyzed (Participants) | 948 | 317
Percentage of participants
  Tetanus: number analyzed (Participants) | 944 | 315
  Tetanus | 74.5 | 81.6
  Diphtheria: number analyzed (Participants) | 945 | 315
  Diphtheria | 83.2 | 84.1
Statistical Analysis 1: Comparison: Adacel Vaccine vs Td Adsorbed Vaccine; Comparison of the anti-tetanus booster response rates between the two groups; Test type: Non-Inferiority — Non-inferiority concluded if the lower limit of the 2-sided 95% CI of the difference of booster response rates between groups is > -10%; Difference (%) in Adacel-Td Adsorbed = -7.12, 95% CI 2-sided [-12.0 to -1.7]
Statistical Analysis 2: Comparison: Adacel Vaccine vs Td Adsorbed Vaccine; Comparison of the anti-diphteria booster response rates between the two groups; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Difference (%) in Adacel-Td Adsorbed = -0.95, 95% CI 2-sided [-5.4 to 4.0]

3. Primary Outcome: Geometric Mean Concentrations (GMC) of Anti Pertussis Antibodies
Description: Anti-Pertussis antibodies (Pertussis toxoid, Filamentous Hemagglutinin (FHA), Pertactin, Fimbriae types 2 and 3) were assessed using an enzyme-linked immunosorbent assay. Anti-pertussis GMCs further to Adacel vaccination was compared to an historical control group with Daptacel (NCT00255047 for pertussis toxoid and PMID 8538705 for FHA, Pertactin and Fimbriae) since Td Adsorbed Vaccine does not contain any pertussis antigens.
Time Frame: 1 month post-booster vaccination
Population: Geometric mean concentrations were assessed in the Per Protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Concentrations (1/dil)
Arm/Group | Adacel Vaccine
Number analyzed (Participants) | 948
Concentrations (1/dil)
  Pertussis Toxoid: number analyzed (Participants) | 935
  Pertussis Toxoid | 102 [94.9 to 110]
  FHA | 209 [200 to 217]
  Pertactin | 318 [302 to 334]
  Fimbriae types 2 and 3 | 745 [711 to 781]
Statistical Analysis 1: Comparison: Adacel Vaccine; Comparison of anti-pertussis toxoid GMCs between Adacel and historical control groups; Test type: Non-Inferiority — Non-inferiority concluded if the lower limit of the 2-sided 95% CI of the ratio of GMCs between groups is > 0.66; GMC ratio (Adacel/Historical Control) = 1.04, 95% CI 2-sided [0.92 to 1.18]
Statistical Analysis 2: Comparison: Adacel Vaccine; Comparison of the anti-FHA GMCs between Adacel and historical Control groups; Test type: Non-Inferiority — Non-inferiority concluded if the lower limit of the 2-sided 95% CI of the ratio of GMCs between groups is > 0.66; GMC Ratio (Adacel/Historical Control) = 5.22, 95% CI 2-sided [4.51 to 6.05]
Statistical Analysis 3: Comparison: Adacel Vaccine; Comparison of the anti-Pertactin GMCs between Adacel and historical Control groups; Test type: Non-Inferiority — Non-inferiority concluded if the lower limit of the 2-sided 95% CI of the ratio of GMCs between groups is > 0.66; GMC Ratio (Adacel/Historical Control) = 2.94, 95% CI 2-sided [2.46 to 3.51]
Statistical Analysis 4: Comparison: Adacel Vaccine; Comparison of the post-vaccination anti-Fimbriae (types 2 and 3) GMCs between Adacel and historical Control groups; Test type: Non-Inferiority — Non-inferiority concluded if the lower limit of the 2-sided 95% CI of the ratio of GMCs between groups is > 0.66; GMC Ratio (Adacel/Historical Control) = 2.18, 95% CI 2-sided [1.84 to 2.60]

4. Primary Outcome: Percentage of Subjects With Pertussis Antigen Booster Response
Description: Anti-Pertussis antibodies (Pertussis toxoid, Filamentous Hemagglutinin [FHA], Pertactin, Fimbriae (types 2 and 3) were assessed using an enzyme-linked immunosorbent assay. Booster response is defined as a minimum rise in antibody concentration from pre- to post-vaccination. The minimum rise is at least 2 times if the pre-vaccination concentration is above the cutoff value, or at least 4 times if it is at or below the cutoff value.
  Anti-pertussis toxoid booster response rates further to Adacel vaccination was compared to an expected booster rates based on study Td506 (PMID 15933223) since Td Adsorbed Vaccine does not contain any pertussis antigens.
Time Frame: 1 month post-booster vaccination
Population: Booster response rate was assessed in the Per protocol analysis set
Measure: Number; unit: Percentage of subjects
Arm/Group | Adacel Vaccine
Number analyzed (Participants) | 948
Percentage of subjects
  Pertussis Toxoid: number analyzed (Participants) | 894
  Pertussis Toxoid | 77.5
  FHA: number analyzed (Participants) | 945
  FHA | 68.9
  Pertactin: number analyzed (Participants) | 945
  Pertactin | 65.3
  Fimbriae (types 2 and 3): number analyzed (Participants) | 945
  Fimbriae (types 2 and 3) | 56.8
Statistical Analysis 1: Comparison: Adacel Vaccine; comparison of anti-pertussis toxoid booster response rates was performed between the Adacel and historical groups; Test type: Non-Inferiority — Non-inferiority concluded if the lower limit of the 2-sided 95% CI of the difference of booster response rates between groups is > -10%; Difference (%) Adacel-Expected Booster = 16.12, 95% CI 2-sided [13.27 to 18.73]
Statistical Analysis 2: Comparison: Adacel Vaccine; Comparison of the anti-FHA booster response rates between the Adacel and historical groups; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Difference (%) Adacel-Expected Booster = -4.21, 95% CI 2-sided [-7.23 to -1.34]
Statistical Analysis 3: Comparison: Adacel Vaccine; Comparison of the anti-Pertactin booster response rates between Adacel and historical groups; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; Difference (%) Adacel-Expected Booster = -18.61, 95% CI 2-sided [-21.7 to -15.6]
Statistical Analysis 4: Comparison: Adacel Vaccine; Comparison of the anti-Fimbriae (types 2 and 3) booster response rates between Adacel and historical groups; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; Difference (%) Adacel-Expected Booster = -19.07, 95% CI 2-sided [-22.3 to -16.0]

5. Secondary Outcome: Percentage of Participants Reporting a Solicited Injection Site or Systemic Reactions
Description: Injection site reactions: Pain, Erythema, and Swelling. Systemic reactions: Fever (Temperature), Headache, Malaise, and Myalgia. Grade 3 Injection site reactions: Pain, Significant, prevents daily activity. Erythema and Swelling, >100 mm. Grade 3 Systemic reactions: Fever, ≥39°C or ≥102.1 F; Headache, Malaise, and Myalgia, Significant; prevents daily activity.
Time Frame: Day 0 up to Day 7 post-vaccination
Population: Solicited injection site and systemic reactions were assessed in the Safety Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | Adacel Vaccine | Td Adsorbed Vaccine
Number analyzed (Participants) | 999 | 328
Percentage of participants
  Any Injection site Pain: number analyzed (Participants) | 982 | 325
  Any Injection site Pain | 87.1 | 87.4
  Grade 3 Injection site Pain: number analyzed (Participants) | 982 | 325
  Grade 3 Injection site Pain | 3.6 | 2.8
  Any Injection site Erythema: number analyzed (Participants) | 982 | 325
  Any Injection site Erythema | 6.4 | 5.5
  Grade 3 Injection site Erythema: number analyzed (Participants) | 982 | 325
  Grade 3 Injection site Erythema | 0.2 | 0
  Any Injection site Swelling: number analyzed (Participants) | 981 | 325
  Any Injection site Swelling | 6.9 | 8.0
  Grade 3 Injection site Swelling: number analyzed (Participants) | 981 | 325
  Grade 3 Injection site Swelling | 0.3 | 0
  Any Fever: number analyzed (Participants) | 978 | 325
  Any Fever | 0.9 | 1.8
  Grade 3 Fever: number analyzed (Participants) | 978 | 325
  Grade 3 Fever | 0.2 | 0.3
  Any Headache: number analyzed (Participants) | 982 | 325
  Any Headache | 41.4 | 39.1
  Grade 3 Headache: number analyzed (Participants) | 982 | 325
  Grade 3 Headache | 2.6 | 4.0
  Any Malaise: number analyzed (Participants) | 982 | 325
  Any Malaise | 33.3 | 30.8
  Grade 3 Malaise: number analyzed (Participants) | 982 | 325
  Grade 3 Malaise | 3.0 | 3.7
  Any Myalgia: number analyzed (Participants) | 982 | 325
  Any Myalgia | 58.1 | 58.2
  Grade 3 Myalgia: number analyzed (Participants) | 982 | 325
  Grade 3 Myalgia | 3.0 | 3.1

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Day 0 up to 1 month post-booster vaccination.
Description: Adverse Events were assessed in the Safety Analysis Set
Arm/Group | Adacel Vaccine | Td Adsorbed Vaccine
All-Cause Mortality (participants affected / at risk) | 0/999 | 0/328
Serious Adverse Events (participants affected / at risk) | 8/999 | 1/328
Other Adverse Events (participants affected / at risk) | 855/999 | 284/328
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adacel Vaccine (N=999) | Td Adsorbed Vaccine (N=328)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Abortion spontaneous (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tonsillar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adacel Vaccine (N=999) | Td Adsorbed Vaccine (N=328)
Injection site Pain (General disorders) | 855 (855) | 284 (284)
Injection site Erythema (General disorders) | 63 (63) | 18 (18)
Injection site Swelling (General disorders) | 68 (68) | 26 (26)
Headache (Nervous system disorders) | 407 (407) | 127 (127)
Malaise (General disorders) | 327 (327) | 100 (100)
Myalgia (Musculoskeletal and connective tissue disorders) | 571 (571) | 189 (189)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications